CLINICAL TRIAL: NCT05745545
Title: A Single-center, Randomized, Blinded, Placebo-controlled Clinical Trial to Evaluate the Protective Efficacy, Safety and Immunogenicity of One Dose of the SARS-CoV-2 Variant (Omicron BA.5) mRNA Vaccine in People Aged 18 Years and Older Who Had Received Two or Three Doses of Inactivated COVID-19 Vaccine
Brief Title: Clinical Trial of COVID-19 Vaccine（SARS-CoV-2 Variant(Omicron BA.5) mRNA Vaccine） in Participants Aged 18 Years and Over
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other); Ningbo Rongan Biological Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LVRNA012-IIT-04
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — mRNA Vaccines; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SARS-CoV-2 Variant (Omicron BA.5) mRNA vaccine (Experimental)
  Interventions: Biological: SARS-CoV-2 Variant (Omicron BA.5) mRNA vaccine
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline solution

INTERVENTIONS:
Biological: SARS-CoV-2 Variant (Omicron BA.5) mRNA vaccine — One dose was administered by intramuscular injection, 100μg，1.0ml/dose
  Arms: SARS-CoV-2 Variant (Omicron BA.5) mRNA vaccine
Drug: Saline solution — One dose was administered by intramuscular injection, 0.5ml/vial
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, blinded, placebo-controlled clinical trial to evaluate the protective efficacy, safety and immunogenicity of one dose of the SARS-CoV-2 variant (Omicron BA.5) mRNA vaccine in people aged 18 years and older who had received two or three doses of inactivated COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female adults aged 18 and above who can provide identification;
2. Know the contents of the informed consent form and the situation of the vaccination, sign the informed consent form voluntarily, and have the ability to use the thermometer, scale and fill in the diary card and contact card as required;
3. Ability to communicate well with researchers, understand and comply with the requirements of the study;
4. Two or three doses of COVID-19 inactivated vaccine have been completed and ≥6 months have passed since the last dose of COVID-19 inactivated vaccine;
5. Healthy subjects or subjects with mild underlying diseases [stable condition with no worsening condition (no need for hospitalization or no major adjustment in treatment regimen, etc.) for at least 3 months prior to inclusion in the study];
6. Women who are not possibility to have children (amenorrhea for at least 1 year or surgical sterilization with medical records) or who are known not to be pregnant or lactating and who have used effective contraception for nearly 14 days before vaccination (e.g., Intrauterine or implantable contraceptive devices,oral contraceptives, injected or embedded contraceptives, slow-release topical contraceptives, intrauterine devices (IUD), condoms (male), diaphragm, cervical cap, etc.) (provide negative proof of pregnancy within 48 hours);
7. SARS-CoV-2 etiology test (RT-PCR) was negative within 48 hours.

Exclusion Criteria:

1. Abnormal vital signs that are clinically significant (e.g. abnormal controlled blood pressure);
2. Have been infected with COVID-19 or used any COVID-19 prophylactic medication other than 3 doses of COVID-19 inactivated vaccine within the last 6 months (for example, a history of any other non-COVID-19 inactivated vaccine on or off the market, or 1 or 4 doses of COVID-19 inactivated vaccine);
3. History of severe acute respiratory syndrome (SARS), Middle East Respiratory Syndrome (MERS) and other human coronavirus infection or disease history;
4. Axillary temperature ≥37.3℃ or fever within 24 hours on the day of vaccination (axillary temperature ≥37.3℃/ mouth temperature ≥37.5℃);
5. A history of severe allergic reactions or allergic reactions to vaccines or drugs, such as urticaria, severe eczema, dyspnea, laryngeal edema, angioneurotic edema, etc.;
6. Vaccination of any vaccine within 28 days prior to study vaccination;
7. Enrolled in a clinical study of another drug within 28 days before vaccination or planned to participate in a clinical study of another drug within 6 months after vaccination;
8. Have a genetic tendency to bleed or abnormal coagulation function (e.g. cytokine deficiency, coagulation disorder or thrombocytopenia), or a history of severe bleeding;
9. A known history or diagnosis of a disease affecting immune system function, such as cancer (other than basal cell carcinoma of the skin), congenital or acquired immunodeficiency (e.g., HIV infection), uncontrolled autoimmune disease, etc.;
10. Asplenia or functional asplenia;
11. Long-term use (continuous use ≥14 days) of immunosuppressants or other immunomodulatory drugs (e.g., cortisol: prednisone or similar drugs) within 6 months prior to study vaccination; Interferon, etc.), but topical use (such as ointments, eye drops, inhalants or nasal sprays) is permitted, and the dose of topical use shall not exceed that recommended in the instructions;
12. Received immunoglobulin and/or blood products within 3 months prior to study vaccination;
13. Suspected or known alcohol dependence or drug abuse;
14. Other factors considered inappropriate to be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Person-year incidence of symptomatic COVID-19 of any severity among persons 18 years of age and older who had received 2 or 3 doses of inactivated COVID-19 vaccine | 14 days after vaccination or placebo
  Person-year incidence of symptomatic COVID-19 of any severity 14 days after vaccination (≥D14) with a booster dose of study vaccine or placebo among persons 18 years of age and older who had received 2 or 3 doses of inactivated COVID-19 vaccine

SECONDARY OUTCOMES:
Person-year incidence of severe and critical COVID-19 in persons aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine | 14 days after vaccination or placebo
  Person-year incidence of severe and critical COVID-19 after 14 days (≥D14) after booster immunization with 1 dose of study vaccine or placebo in persons aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine
Person-year incidence of COVID-19 resulting in death in persons aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine | 14 days after vaccination or placebo
  Person-year incidence of COVID-19 resulting in death 14 days (≥D14) after booster vaccination with 1 dose of study vaccine or placebo in persons aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine
Person-year incidence of symptomatic COVID-19 of any severity among persons aged 18-59 years and ≥60 years who had received 2 or 3 doses of inactivated COVID-19 vaccine | 14 days after vaccination or placebo
  Person-year incidence of symptomatic COVID-19 of any severity 14 days (≥D14) after booster immunization with 1 dose of study vaccine or placebo among persons aged 18-59 years and ≥60 years who had received 2 or 3 doses of inactivated COVID-19 vaccine
GMT of true virus neutralizing antibodies against the current major circulating strain of SARS-CoV-2 in subjects in the immunization subgroup | 7 days, 14 days, 28 days, 3 months, and 6 months after vaccination or placebo
  In the immunization subgroup, true virus neutralizing antibodies GMT against the current major circulating strain of SARS-CoV-2 were detected 7 days, 14 days, 28 days, 3 months, and 6 months after receiving one dose of study vaccine or placebo
GMI of true virus neutralizing antibodies against the current major circulating strain of SARS-CoV-2 in subjects in the immunization subgroup | 7 days, 14 days, 28 days, 3 months, and 6 months after vaccination or placebo
  In the immunization subgroup, true virus neutralizing antibodies GMI against the current major circulating strain of SARS-CoV-2 were detected 7 days, 14 days, 28 days, 3 months, and 6 months after receiving one dose of study vaccine or placebo
SCR of true virus neutralizing antibodies against the current major circulating strain of SARS-CoV-2 in subjects in the immunization subgroup | 7 days, 14 days, 28 days, 3 months, and 6 months after vaccination or placebo
  In the immunization subgroup, true virus neutralizing antibodies SCR against the current major circulating strain of SARS-CoV-2 were detected 7 days, 14 days, 28 days, 3 months, and 6 months after receiving one dose of study vaccine or placebo
GMT of S protein IgG against the current major circulating strain of SARS-CoV-2 in the immunization subgroup | 7 days, 14 days, 28 days, 3 months, and 6 months after vaccination or placebo
  GMT of S protein IgG against the current major circulating strain of SARS-CoV-2 7 days, 14 days, 28 days, 3 months, and 6 months after receiving one dose of study vaccine or placebo in the immunization subgroup
GMI of S protein IgG against the current major circulating strain of SARS-CoV-2 in the immunization subgroup | 7 days, 14 days, 28 days, 3 months, and 6 months after vaccination or placebo
  GMI of S protein IgG against the current major circulating strain of SARS-CoV-2 7 days, 14 days, 28 days, 3 months, and 6 months after receiving one dose of study vaccine or placebo in the immunization subgroup
SCR of S protein IgG against the current major circulating strain of SARS-CoV-2 in the immunization subgroup | 7 days, 14 days, 28 days, 3 months, and 6 months after vaccination or placebo
  SCR of S protein IgG against the current major circulating strain of SARS-CoV-2 7 days, 14 days, 28 days, 3 months, and 6 months after receiving one dose of study vaccine or placebo in the immunization subgroup
Incidence of adverse events in people aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine | 30 minutes, 0-14 days and 0-28 days after vaccination or placebo
  Incidence of adverse events at 30 minutes, 0-14 days and 0-28 days after booster vaccination of 1 dose of study vaccine or placebo in people aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine
Incidence of serious adverse events (SAE) in people aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine | within 6 months after vaccination or placebo
  Incidence of serious adverse events (SAE) within 6 months after booster immunization with 1 dose of study vaccine or placebo in people aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine
Incidence of AESI in people aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine | within 6 months after vaccination or placebo
  Incidence of AESI within 6 months after booster immunization with 1 dose of study vaccine or placebo in people aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine
Pregnancy events among persons aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine | within 6 months after vaccination or placebo
  Pregnancy events within 6 months after booster vaccination with 1 dose of study vaccine or placebo (including: pregnancy outcomes, delivery characteristics, delivery of newborns, and growth and development within 1 month after birth) among persons aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine

OTHER OUTCOMES:
Person-year incidence of COVID-19 of any severity in persons aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine | 7 days after vaccination or placebo
  Person-year incidence of COVID-19 of any severity 7 days after vaccination (≥D7) with a booster dose of study vaccine or placebo in persons aged 18 years and older who had received 2 or 3 doses of inactivated COVID-19 vaccine
Immune subgroup: viral antigen IL-2 levels | 7 days, 14 days, 28 days and 3 months after vaccination or placebo
  Immune subgroup: viral antigen IL-2 levels at 7 days, 14 days, 28 days and 3 months after vaccination (ELISpot assay)
Immune subgroup: viral antigen IL-4 levels | 7 days, 14 days, 28 days and 3 months after vaccination or placebo
  Immune subgroup: viral antigen IL-4 levels at 7 days, 14 days, 28 days and 3 months after vaccination (ELISpot assay)
Immune subgroup: viral antigen IL-13 levels | 7 days, 14 days, 28 days and 3 months after vaccination or placebo
  Immune subgroup: viral antigen IL-13 levels at 7 days, 14 days, 28 days and 3 months after vaccination (ELISpot assay)
Immune subgroup: viral antigen IFN-γ cytokine levels | 7 days, 14 days, 28 days and 3 months after vaccination or placebo
  Immune subgroup: viral antigen IFN-γ cytokine levels at 7 days, 14 days, 28 days and 3 months after vaccination (ELISpot assay)
The correlation between neutralizing antibodies, S-protein IgG antibodies and/or cellular immunoassay data protective efficacy | 6 months after vaccination or placebo
  To explore the correlation between neutralizing antibodies, S-protein IgG antibodies and/or cellular immunoassay data after vaccination and vaccine protective efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Qiang Wu, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui, China

REFERENCES:
- [Derived] Vetter VM, Kurth T, Konigorski S. Evaluation of easy-to-implement anti-stress interventions in a series of N-of-1 trials: study protocol of the anti-stress intervention among physicians study. Front Psychiatry. 2024 Aug 23;15:1420097. doi: 10.3389/fpsyt.2024.1420097. eCollection 2024. PMID 39247614
- [Derived] Emadi Torghabeh A, Aledavood SA, Soltani E, Akbari Oryani M, Akhlaghi S, Hosseini S, Fani Pakdel A, Taghizadeh Kermani A, Anvari K, Shahidsales S, Bahadorian S, Mashreghi Moghaddam S. Pathologic response evaluation of localized or locally advanced esophageal carcinoma to induction chemotherapy followed by preoperative concurrent chemotherapy and hypofractionated radiotherapy: a clinical trial. Front Oncol. 2024 Aug 19;14:1439730. doi: 10.3389/fonc.2024.1439730. eCollection 2024. PMID 39224811
- [Derived] Zhou H, Zheng H, Peng Y, Su Y, Yu X, Wang W, Li S, Ding Y, Jiao S, Wang Y, Zhu X, Luo L, Dong Z, Liu L, Zhang F, Wu Q, Li J, Zhu F. Efficacy, safety, and immunogenicity of SARS-CoV-2 mRNA vaccine (Omicron BA.5) LVRNA012: a randomized, double-blind, placebo-controlled phase 3 trial. Front Immunol. 2024 Jun 6;15:1407826. doi: 10.3389/fimmu.2024.1407826. eCollection 2024. PMID 38903523